CLINICAL TRIAL: NCT06261541
Title: Clinical Investigation to Validate the Safety and Performance of the ABLE Exoskeleton Device for Individuals With Multiple Sclerosis in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: Fundación Esclerosis Múltiple Madrid (FEMM) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABLEexoMS
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Lower-limb exoskeleton; Gait training
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait training with exoskeleton (Experimental): Participants with MS will undergo a training program with the ABLE Exoskeleton device: a total of 10 sessions, distributed 1-2 sessions/week for up to 11 weeks.
  Interventions: Device: ABLE Exoskeleton

INTERVENTIONS:
Device: ABLE Exoskeleton — Participants with MS will undergo a training program with the ABLE Exoskeleton device: a total of 10 sessions, distributed 1-2 sessions/week for up to 11 weeks.

SUMMARY:
The primary objective of the study is to validate the safety and performance of the ABLE Exoskeleton device in people with multiple sclerosis during a 10-session gait training program in a clinical setting. Furthermore, the potential effects of the training on walking, and balance function, general health status, user satisfaction, and quality of life will be assessed.

DETAILED DESCRIPTION:
This is a pre-post, single-center, quasi-experimental study with an estimated duration of 4 months since the approval date. The study will be conducted at the Fundación Esclerosis Múltiple de Madrid (FEMM), where a minimum of 20 participants are expected to be recruited over a maximum period of 2 months since the approval date.

After obtaining informed consent, through the Patient Information Sheet and the Informed Consent Form, the selection of the participants will be carried out to determine their inclusion in the study. Subjects who do not meet all the inclusion and exclusion criteria during the screening visit will be excluded from the study. At the latest, one week after the screening visit, the participants will undergo a preliminary assessment without the medical device.

Participants will undergo a 10-session training program with the ABLE Exoskeleton device for a maximum duration of 11 weeks. Sessions will be conducted 1 to 2 times per week, depending on the participant's availability. Each session will last approximately 60 minutes. During the training period, session data will be taken to assess the safety and clinical performance of the device. At the latest, one week after the last training session, a post-training assessment will be performed. Finally, two weeks after the last training session, a follow-up assessment will be made to the participants via a telephone call to review any adverse events (AE) reported between the end of the training and the follow-up.

This is the first study investigating the use of the ABLE Exoskeleton in people with MS, therefore the primary hypothesis of this study is that the ABLE Exoskeleton is safe and has adequate performance for the intended MS population in a clinical setting. The secondary hypothesis is that the device will have a positive impact on the muscular strength, spasticity, perceived rate of exertion, mobility, satisfaction, and quality of life of the study participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age.
* Diagnosed with MS.
* Currently receiving treatment as an inpatient or outpatient at one of the investigational site.
* Ability to give informed consent.

Exclusion Criteria:

* Significant osteoporosis that may increase the risk of fracture.
* Unresolved fractures in the pelvis or extremities, or history of fragility fractures in the lower extremities in the last 2 years.
* Spinal instability (or spinal orthoses, unless authorized by a physician).
* Severe spasticity: Level 4 on the Modified Ashworth Scale.
* Orthostatic hypotension. Inability to tolerate a minimum of 30 minutes of standing.
* Uncontrolled autonomic dysreflexia.
* Medically unstable
* Unstable cardiovascular system (CVS), hemodynamic instability, untreated hypertension (SBP>140, DBP>90 mmHg), unresolved deep venous thrombosis (DVT).
* Serious comorbidities, including any condition that a physician deems inappropriate for use of the ABLE Exoskeleton or to complete participation in the study.
* Skin integrity problems on the contact surfaces of the device or that would prevent sitting.
* Grade I or higher on EPUAP (European Pressure Ulcer Advisory Panel, 2019) on areas that will be in contact with the exoskeleton.
* Colostomy.
* Anthropometric measurements outside the values compatible with ABLE Exoskeleton. In particular, height not between 1.5-1.9 m, or weight over 100 kg.
* Anatomical constraints (such as eg length differences, users unable to position themselves inside the device) that are incompatible with the device.
* Restrictions in range of motion that prevent normal gait from being achieved or preventing the completion of a normal transition from sitting to standing or standing to sitting.
* Heterotopic ossification
* Known pregnancy or breastfeeding
* Cognitive impairment that results in the inability to follow simple instructions, particularly psychological or cognitive problems that do not allow a participant to follow study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Number and type of device-related Adverse Events | Up to 16 weeks
  To assess safety, the number of Severe Adverse Events (SAE), Adverse Events (AE) and drop-outs due to the device will be assessed and reported.
Level of Assistance (LoA) to don/doff the device | Up to 11 weeks
  Level of Assistance (LoA) to don/doff the device will be measured in every session. The level of assistance will be measured using a 6-item scale, from Total assistance to Independence, with Independence being the best outcome possible. Different assistance levels are defined taking into account the degree of participation of both the participant and the therapist on performing the activity.
Time taken to don/doff the device | Up to 11 weeks
  The time taken to don/doff the device will be measured in every session. Time will be measured in minutes and seconds for each activity. Donning time will start from the moment the participant is ready to transfer into the device until all the straps and clips are correctly tightened. Doffing time will start from the moment the participant starts taking off the device until they have completely removed it.
Level of Assistance (LoA) to complete therapy activity tasks | Up to 11 weeks
  Four therapy activity tasks will be attempted every session by the participant. The therapist will record the level of assistance required to complete each task during the session, using a 6-item scale, from Total assistance to Independence, with Independence being the best outcome possible. The tasks are the following: sit-to-stand, walk 10 meters, turn 180 degrees, and stand-to-sit.
Time spent upright and time spent walking | Up to 11 weeks
  In each training session, the time spent upright (in minutes) and the time spent walking (in minutes) with the device will be automatically measured and registered by the device.
Number of steps walked | Up to 11 weeks
  In each session, the number of steps taken (step count) with the device will be automatically measured and registered by the device.
Distance walked | Up to 11 weeks
  In each session, the distance walked (in meters) with the device will be automatically measured and registered by the device.

SECONDARY OUTCOMES:
Timed 25-Feet Walk test (T25FW) | Up to 11 weeks
  The Timed 25-Foot Walk (T25FW) test measures the time a person needs to walk 25 feet. This test will be performed in the pre-post evaluations without the device to assess the change in the walking function after the training.
Ambulation Index (AI) | Up to 11 weeks
  The Ambulation Index (AI) is a rating scale that assesses mobility based on time and degree of assistance required when walking 25 feet as quickly as possible but safely. Scores range from 0 (asymptomatic and fully active) to 10 (bedridden). This test will be performed in the pre-post evaluations without the device to assess the change in the walking function after the training.
6-Minute Walk Test (6MWT) | Up to 11 weeks
  The 6-Minute Walk Test (6MWT) measures the distance a person can walk in 6 minutes. This test will be performed in the pre-post evaluations without the device to assess the change in the walking function after the training.
Timed Up-and-Go test (TUG) | Up to 11 weeks
  The Timed Up-and-Go Test (TUG) measures the time it takes a person to get up from a chair, walk 3 meters, turn around, and sit down again. This test will be performed in the pre-post evaluations without the device to assess the change in the walking function after the training.
Trunk Impairment Scale (TIS) | Up to 11 weeks
  The Trunk Impairment Scale (TIS) measures the motor impairment of the trunk through the evaluation of static and dynamic sitting balance as well as coordination of trunk movement. The total score ranges from 0 (minimal performance) to 23 (perfect performance). This test will be performed in the pre-post evaluations without the device to assess the change in the trunk impairment after training.
Lower extremity muscle strenght | Up to 11 weeks
  The Daniels Muscle Testing scale will be used to measure the strength of muscles in the lower extremities in the pre-post evaluations to assess motor function after the training. Scores range from 0 (absence of muscle activity) to 5 (normal muscle activity).
Modified Ashworth Scale (MAS) | Up to 11 weeks
  The Modified Ashworth Scale (MAS) measures spasticity in patients with lesions to the central nervous system. The scale assigns a grade of spasticity from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). It will be evaluated in the pre-post evaluations without the device to assess the change in the spasticity after training.
Borg Rating of Perceived Exertion | Up to 11 weeks
  The Borg Rating of Perceived Exertion (RPE) scale is used to measure a person's perception of their effort and exertion, breathlessness, and fatigue during physical activity. Scores range from 6 (no exertion at all) to 20 (maximal exertion). It will be evaluated in the pre-post evaluations without the device to assess the change in the perceived exertion after the training.
Barthel Index (BI) score | Up to 11 weeks
  The Barthel Index (BI) will be used to assess the participants' ability to perform mobility and self-care activities of daily living (ADL). The total score ranges from 0 (total dependency) to 100 (independency). It will be evaluated in the pre-post evaluations without the device to assess the change in the independence to perform ADL after the training.
Modified Fatigue Impact Scale (MFIS) score | Up to 11 weeks
  The Modified Fatigue Impact Scale (MFIS) provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning in persons with multiple sclerosis. The total score ranges from 0 to 84, with higher scores meaning a higher impact of fatigue. It will be evaluated in the pre-post evaluations without the device to assess the change in the fatigue after the training.
Multiple Sclerosis Quality of Life-54 (MSQoL-54) | Up to 11 weeks
  The Multiple Sclerosis Quality of Life-54 (MSQoL-54) is a multidimensional health-related quality of life (QoL) measure that combines both generic and MS-specific items into a single instrument. There is no single overall score for the MSQoL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores. The higher the score, the best the outcome. It will be evaluated in the pre-post evaluations without the device to assess the change in the QoL after the training.
Psychosocial Impact of Assistive Devices Scale (PIADS) score | Up to 11 weeks
  The Psychosocial Impact of Assistive Devices Scale (PIADS) is a 26-item, self-reported questionnaire that provides a measure of user perception and other psychological factors associated with assistive technology devices. Scores range from -78 (maximum negative impact) to +78 (maximum positive impact). It will be used to assess the effects of the ABLE Exoskeleton on functional independence, well-being, and quality of life of participants after the training program experience.
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) score | Up to 11 weeks
  The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) is a 12-item outcome measure that assesses user satisfaction with two components (Device and Services) using a 5-point scale ranging from 1 (not satisfied) to 5 (very satisfied). Only the 8 items referred to the device will be evaluated to measure user satisfaction from participants and therapists with the ABLE Exoskeleton after the training program experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Esclerosis Múltiple Madrid (FEMM), Madrid, Spain